CLINICAL TRIAL: NCT00054678
Title: A Phase I, Open-Label, Non-Randomized, Dose Escalation, Multi Center Study to Assess the Safety and Cardiovascular Effects of Autologous Skeletal Myoblast Implantation by a Transendocardial Catheter Delivery System in Congestive Heart Failure Patients Post Myocardial Infarction(s) With Previous Placement of ICD
Brief Title: MYOHEART™ (Myogenesis Heart Efficiency and Regeneration Trial)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bioheart, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMI-US-01-002; Version G
Record Dates: First submitted 2003-02-06; First posted 2003-02-07 (Estimated); Last update posted 2007-10-15 (Estimated); Status verified 2007-10

CONDITIONS: Congestive Heart Failure; Coronary Artery Disease; Myocardial Infarction
Keywords: Myocardial infarction; Heart disease; Endoventricular; Cardiovascular; Interventional; ICD; Heart failure; Implantable Cardioverter Defibrillator
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease; Myocardial Infarction; Heart Diseases

INTERVENTIONS:
Drug: MyoCell™
Device: MyoCath™

SUMMARY:
The MyoCell™ implantation using the MyoCath™ delivery catheter system may have the potential to add a new dimension to the management of post-infarct deterioration of cardiac function in subjects with congestive heart failure. Based on pre-clinical studies, implantation of autologous skeletal myoblasts may lead to replacement of non-functioning myocardial scar with functioning muscle and improvement in myocardial performance. Preliminary data in human subjects suggest skeletal myoblast implantation at the time of CABG may lead to the same effects. In principal, myoblast implantation by catheter delivery may offer the same therapeutic benefit. The present clinical study is to be conducted primarily to evaluate the safety of MyoCell™ implantation using the MyoCath™ delivery system and secondarily to evaluate the effect on regional myocardial function post treatment.

DETAILED DESCRIPTION:
A very promising approach to reversal or stabilization of the post-infarct remodeling process is the direct injection of regenerative cells into the myocardial infarct scar. Such cell-based therapy for cardiac repair is called "cellular cardiomyoplasty".

The MyoCell™ implantation using the MyoCath™ delivery catheter system may have the potential to add a new dimension to the management of post-infarct deterioration of cardiac function in subjects with congestive heart failure. MyoCath™ is Bioheart's proprietary catheter delivery system being developed by Bioheart to facilitate MyoCell™ delivery into the myocardium via the retrograde catheterization of the left ventricular cavity. Based on pre-clinical studies, implantation of autologous skeletal myoblasts may lead to replacement of non-functioning myocardial scar with functioning muscle and improvement in myocardial performance. Preliminary data in human subjects suggest skeletal myoblast implantation at the time of CABG or via the endoventricular approach may lead to the same effects. In principle, myoblast implantation by catheter delivery may offer the same therapeutic benefit.

The present clinical study is to be conducted primarily to:

1. Assess the safety and effect on myocardial function of MyoCell™ (autologous skeletal myoblast) using a dose escalation methodology following implantation into myocardial scar tissue of subjects with congestive heart failure who have experienced previous myocardial infarction(s) and have had an implantable cardioverter defibrillator (ICD) previously implanted. Safety endpoints will be the evaluation of the nature and frequency of Adverse Events during the 12-month period following MyoCell™ treatment.
2. To assess the safety and feasibility of using the transendocardial injection catheter (MyoCath™) as a system for delivering MyoCell™ into myocardial scar tissue of subjects with congestive heart failure who have experienced previous myocardial infarction(s) and have an implantable cardioverter defibrillator (ICD) previously implanted. Catheter performance will be assessed at the time of the implantation using clinical evaluation questionnaires. Safety endpoints will be the evaluation of the nature and frequency of Adverse Events from the time of implantation to the Day 14 follow-up visit.

If a patient meets the baseline enrollment criteria, approximately 5-10 grams of skeletal muscle is obtained from the subject's leg muscle for myoblast isolation and expansion in vitro (MyoCell™) at a specified off site cGMP culture laboratory. The expanded myoblast cells, MyoCell™ will be implanted into the akinetic myocardial scar in the region of a previous infarct utilizing Bioheart's MyoCath™ transendocardial delivery catheter system. The MyoCath™ endoventricular device is expected to deliver the MyoCell™ autologous skeletal myoblast cells into the scarred myocardial region by steering a catheter which contains a retractable hypodermic needle to the targeted sites for implantation.

This will be a dose escalation study with 4 cohort groups consisting of 5 patients each. A report of the 1 month safety data from each cohort will be presented to the Data Safety Monitoring Board for permission to go to the next higher dosage. In the first cohort of this dose escalation study, 2 injections will be performed; for the second cohort, 6 injections; for the third cohort, 18 injections; and for the fourth cohort, 27 injections, depending on the size of the infarct scar, so as to inject the entire myocardial infarct scar akinetic area.

The entire study is expected to be completed during the first half of 2007, including completed enrollment as well as 12-month follow-up of the last subject.

ELIGIBILITY:
Patients who meet all of the following inclusion criteria and none of the exclusion criteria will be enrolled in this clinical study.

Inclusion Criteria:

* Defined region of myocardial dysfunction related to previous myocardial infarction(s) involving the anterior, lateral, posterior or inferior walls, > 12 weeks (84 days) old at the scheduled time of MyoCell™ implantation
* Patients who have had prior placement of an Implantable Cardioverter Defibrillator (ICD) which must be in place at least one month (30 days) prior to MyoCell™ implantation
* New York Heart Association (NYHA) Symptom Class II or III on optimal medical therapy
* Age > 30 and < 80 years old
* Need for revascularization has been ruled out by coronary angiogram or noninvasive stress testing within six months (180 days) of screening
* Able to undergo surgical biopsy of the skeletal muscle and successful culture of the harvested myoblasts Target region wall thickness > 6 mm by Echocardiography
* Left ventricular ejection fraction > 20% and < 40% by Radionuclide Ventriculography or Left Ventricular Angiography at screening
* Able to give written informed consent
* Able to walk a minimum distance of 300 meters during the 6-minute walk test

Exclusion Criteria:

* Myocardial infarction within 12 weeks (84 days) prior to investigational procedure
* New York Heart Association Symptom Class I or IV
* Coronary Artery Bypass Grafting (CABG) within 3 months (90 days) prior to scheduled MyoCell™ implantation
* Percutaneous Coronary Intervention (PCI) within 6 months (180 days) prior to MyoCell™ implantation
* Canadian Heart Classification of angina > Class II or unstable angina
* Any cardiac valve replacement
* Heart failure secondary to valvular disease
* Aortic stenosis greater than mild degree
* Left ventricular or atrial mural thrombus
* Chronic pulmonary disease
* Atherosclerosis and/or tortuosity of the aorta, iliac or femoral arteries of a degree which, in the judgment of the principal investigator, would impede or preclude the safe retrograde passage of the 8FR MyoCath™ delivery catheter
* History of severe radiocontrast reaction
* Known sensitivity to gentamicin sulfate and/or amphotericin-B
* Previous angiogenic therapy and/or myocardial laser therapy
* Exposure to any investigational drug or procedure within 1 month prior to study entry
* The use or expected use of antineoplastic drugs or history of cancer within 5 years, except for basal cell carcinoma of the skin
* Skeletal muscle disease, either primary (i.e., myopathy) or secondary (i.e., ischemic) or any underlying myopathy such as myasthenia gravis, muscular dystrophy, etc. as determined by a board certified pathologist examining sample of patients muscle biopsy
* Serum creatinine > 2.5 mg/dL or end stage renal disease
* Prostate Specific Antigen (PSA) suggestive of carcinoma of the prostate (i.e., > 4.0 ng/mL)
* Carcinoembryonic Antigen (CEA) >5.0 ng/mL or end stage renal disease
* Active infectious disease and/or who are known to have tested positive for HIV, HTLV, HBV-sAg, HCV, CMV and/or syphilis. If the panel includes antibodies to the HBc and HBV-sAg, then an expert will be consulted as to patient eligibility based on the patient's infectious status
* Females who are pregnant or nursing
* Females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Morbid obesity - more than 100 pounds over ideal body weight or Body Mass Index (BMI) > 40
* Any illness which might affect patient's survival over the study 12 month follow-up period*
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* No written Informed Consent or unable to provide informed consent

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-02; Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of Myocel following implantation into myocardial scar tissue of subjects with congestive heart failure who have experienced previous MI.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Sherman, MD, Principal Investigator — Columbia University; Timothy Henry, MD, Principal Investigator — Minneapolis Heart / Abbott Northwestern; Nicolas Chronos, MD, Principal Investigator — St. Joseph Hospital / ACRI; Steven Elliss, MD, Principal Investigator — The Cleveland Clinic; David Holmes, MD, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - SPONSOR: Bioheart, Inc, Sunrise, Florida
  - American CardioVascular Research Institute, Atlanta, Georgia
  - Minneapolis Heart Institute / Abbot Northwestern, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Cleveland Clinic Heart Center, Cleveland, Ohio

REFERENCES:
- See also: Bioheart, Incorporated website — http://www.bioheartinc.com
- See also: American Heart Association — http://www.americanheart.org